CLINICAL TRIAL: NCT03058744
Title: A Phase 1b Open Label, Randomized Study Evaluating the Absorption and Systemic Pharmacokinetics and HPA Axis Suppression Potential of Topically Applied IDP-118 Lotion and HP Monad Lotion in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: Topically Applied IDP-118 Lotion and HP Monad Lotion in Subjects With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V01-118A-501
Record Dates: First submitted 2016-12-21; First posted 2017-02-23 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — halobetasol; Transcriptional Coactivator with PDZ-Binding Motif Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- IDP-118 Lotion (Experimental): 8 Weeks
  Interventions: Drug: IDP-118 Lotion
- HP Monad Lotion (Experimental): 8 Weeks
  Interventions: Drug: HP Monad Lotion
- Ultravate Cream (Active Comparator): 2 Weeks
  Interventions: Drug: Ultravate Cream
- Tazorac Cream (Active Comparator): 4 Weeks
  Interventions: Drug: Tazorac Cream

INTERVENTIONS:
Drug: IDP-118 Lotion — Lotion
  Other Names: Lotion
  Arms: IDP-118 Lotion
Drug: HP Monad Lotion — Lotion
  Other Names: Lotion
  Arms: HP Monad Lotion
Drug: Ultravate Cream — Cream
  Other Names: Ultravate
  Arms: Ultravate Cream
Drug: Tazorac Cream — Cream
  Other Names: Taz
  Arms: Tazorac Cream

SUMMARY:
Suppression Potential of Topically Applied IDP-118 Lotion and HP Monad Lotion in Subjects with Moderate to Severe Plaque Psoriasis.

DETAILED DESCRIPTION:
A Phase 1b Open-Label, Randomized Study Evaluating the Absorption and Systemic Pharmacokinetics and HPA Axis Suppression Potential of Topically Applied IDP-118 Lotion and HP Monad Lotion in Subjects with Moderate to Severe Plaque Psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female of any race, at least 18 years old of age (inclusive)
* Freely provides both written and oral informed consent.
* Has a clinical diagnosis of psoriasis at the Baseline visit with an Investigator's Global Assessment Score of 3 or 4. The face, scalp ,axillae, and intertriginous areas are to be excluded in this calculation.
* Has an area of plaque psoriasis for topical treatment that involves a BSA of at least 20%.
* The willing and able to avoid prolonged exposure of the treatment area to ultraviolet radiation (natural and artificial) for the duration of the study.

Key Exclusion Criteria:

* Has spontaneously improving or rapidly deteriorating plaque psoriasis or postural psoriasis, as determined by the investigator.
* Presents with psoriasis that was treated with prescription medication and failed to respond to presents).
* Has a history of adrenal disease.
* Presents with any other concurrent skin conditions that could interfere with the evaluation of the treatment areas, as determined by the investigator.
* Is pregnant, nursing, or planning pregnancy during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Local Skin Reactions (LSRs) | 8 Weeks
  Tolerability will be evaluated through assessment of local signs and symptoms (itching, dryness, burning/stinging) on a scale of non, mild, moderate, and severe.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Mathew, Study Director — Valeant Pharmaceuticals
Locations (12):
- United States (12):
  - Valeant Site 12, Anaheim, California
  - Valeant Site 05, Encino, California
  - Valeant Site 01, San Diego, California
  - Valeant Site 07, Santa Rosa, California
  - Valeant Site 10, Orange Park, Florida
  - Valeant Site 09, Sanford, Florida
  - Valeant Site 08, Atlanta, Georgia
  - Valeant Site 04, Plainfield, Indiana
  - Valeant Site 06, New York, New York
  - Valeant Site 11, Philadelphia, Pennsylvania
  - Valeant Site 03, Austin, Texas
  - Valeant Site 02, Katy, Texas

IPD SHARING:
Plan to Share IPD: Yes